CLINICAL TRIAL: NCT03625908
Title: Optical CoherenCe Tomography-gUided Coronary Intervention in Patients With Complex lesIons: a Randomized Controlled Trial (OCCUPI Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1-2018-0018
Record Dates: First submitted 2018-06-11; First posted 2018-08-10 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Optical coherence tomography; antiplatelet therapy
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients will be assigned by use of OCT-guidance or angiography-guidance for stent implantation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OCT-guided PCI (Active Comparator): Patients will receive PCI under OCT-guidance.
  Interventions: Device: OCT-guided PCI
- Angiography-guided PCI (Active Comparator): Patients will receive PCI under Angiography-guidance.
  Interventions: Device: Angiography-guided PCI

INTERVENTIONS:
Device: OCT-guided PCI — Patients will receive PCI under OCT-guidance. Predefined criteria for optimization of PCI under OCT-guidance will be recommended to achieve as far as possible.
  Arms: OCT-guided PCI
Device: Angiography-guided PCI — Stent optimization using high-pressure non-compliance balloon will be highly recommend. Balloon size would not be less than the stent diameter.
  Arms: Angiography-guided PCI

SUMMARY:
There is no definite conclusive work about the benefit of OCT-guided PCI, which should be determined in complex PCI, assuming better stent optimization by OCT. In the study, we will explore the clinical implication of OCT-guided PCI of complex lesions.

DETAILED DESCRIPTION:
Eligible patients will be randomly assigned to either OCT-guided PCI arm and angiography-guided PCI with routine high pressure NC ballooning arm in 1:1 ratio. Within OCT-guided PCI arm, the use of OCT will be also assigned to full OCT-guidance arm and postprocedural OCT only arm. and comparison of stent implantation with and without preprocedural OCT will be evaluated by postprocedural OCT (OCT-defined stent optimization will be assessed). In angiography-guided PCI arm, PCI for complex lesion will be performed without guidance of intravascular imaging, and routine use of high pressure postdilation with NC balloon will be also recommended. Primary endpoint will be evaluated during 12 months after PCI.

ELIGIBILITY:
Inclusion criteria

* Age 19-85 years
* Patients with ischemic heart diseases (including stable angina, unstable angina and acute myocardial infarction) presented with typical chest pain or objective evidences of myocardial ischemia (positive invasive or non-invasive studies, electrocardiogram (ECG) consistent with ischemia, or elevated cardiac enzymes)
* Complex coronary stenotic lesions (>50% based on visual estimate) considered for coronary revascularization with DES
* Definition of complex lesions (at least one):

  * Acute myocardial infarction
  * Chronic total occlusion
  * Long lesion: expected stent length ≥28mm based on angiographic estimation
  * Calcified lesion
  * Bifurcation (including all techniques, one- or two-stent)
  * Unprotected left main disease
  * Small vessel diseases with reference vessel diameter less than 2.5 mm
  * Intracoronary thrombus visible on the angiography
  * Stent thrombosis
  * In-stent restenosis
  * Bypass graft lesion
* Patients who provide signed informed consent

Exclusion criteria

* Severe hepatic dysfunction (≥3 times normal reference values)
* Significant renal dysfunction (Serum creatinine >2.0 mg/dL)
* Platelet count <100,000 cells/mm3 or >700,000 cells/mm3, a white blood cell count of <3,000 cells/mm3, hemoglobin <8.0 g/dL, or other known bleeding diathesis
* Hemodynamically unstable during procedures or cardiogenic shock
* Pregnant women or women who might be pregnant
* Life expectancy; less than 1 year
* Inability to understand or read the informed content

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1604 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Composite of major adverse cardiac events (MACEs) | 1 year
  Composite of major adverse cardiac events (MACEs) - for comparison between OCT-guided PCI vs. angiography-guided PCI

SECONDARY OUTCOMES:
Each component of MACE | 1 year (except periprocedural MI - within 48 hours)
  MACE = composite of cardiac death, myocardial infarction, stent thrombosis, ischemia-driven target vessel revascularization
Any revascularization | 1 year (except periprocedural MI - within 48 hours)
Target lesion revascularization | 1 year (except periprocedural MI - within 48 hours)
Periprocedural myocardial infarction | 1 year (except periprocedural MI - within 48 hours)
  Periprocedural MI - PCI-related myocardial infarction (>5x or >10x ULN)
Bleeding | 1 year (except periprocedural MI - within 48 hours)
  Bleeding defined by BARC and TIMI criteria
Stroke | 1 year (except periprocedural MI - within 48 hours)
Stent optimization confirmed by OCT | 1 year (except periprocedural MI - within 48 hours)
  The attainment(optimal or acceptable) of criteria regarding stent expansion is strongly recommended. As for the other criteria, further procedures could be decided by the operators' decisions considering the situations.
  1. Stent expansion Optimal - meeting of all criteria Acceptable - meeting of any one criteria 1) MSA≥80% of mean reference lumen area 2) ≥100% of distal reference lumen area 3) MSA of >4.5 mm2 in non-left main lesion
  2. Stent apposition Optimal - acute stent malposition<200μm Acceptable - acute stent malposition<400μm
  3. Edge dissection(Definition of major edge dissection; any one of the followings) 1) ≥60°of the circumference of the vessel at site of dissection 2) Length of dissection ≥3mm 3) Deeper vessel injury(intramural hematoma or penetration to the media or adventitia)
Contrast-induced Nephropathy | 1 year (except periprocedural MI - within 48 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Cardiovascular Center and Cardiovascular Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee YJ, Kim Y, Lee OH, Cho DK, Lee SH, Lee SJ, Lee JY, Kim JW, Kim SM, Hur SH, Heo JH, Jang JY, Koh JS, Won H, Lee JW, Hong SJ, Kim DK, Choe JC, Lee JB, Yang TH, Lee JH, Hong YJ, Ahn JH, Hong SJ, Ahn CM, Kim JS, Ko YG, Choi D, Hong MK, Jang Y, Kim BK, Occupi Investigators OBOT. Optical coherence tomography-guided percutaneous coronary intervention in acute coronary syndrome patients with complex lesions: a subgroup analysis of the randomised OCCUPI Trial. EuroIntervention. 2025 Nov 3;21(21):e1269-e1280. doi: 10.4244/EIJ-D-25-00478. PMID 41489717
- [Derived] Hong SJ, Lee SJ, Lee SH, Lee JY, Cho DK, Kim JW, Kim SM, Hur SH, Heo JH, Jang JY, Koh JS, Won H, Lee JW, Hong SJ, Kim DK, Choe JC, Lee JB, Kim SJ, Yang TH, Lee JH, Hong YJ, Ahn JH, Lee YJ, Ahn CM, Kim JS, Ko YG, Choi D, Hong MK, Jang Y, Kim BK; OCCUPI investigators. Optical coherence tomography-guided versus angiography-guided percutaneous coronary intervention for patients with complex lesions (OCCUPI): an investigator-initiated, multicentre, randomised, open-label, superiority trial in South Korea. Lancet. 2024 Sep 14;404(10457):1029-1039. doi: 10.1016/S0140-6736(24)01454-5. Epub 2024 Sep 2. PMID 39236729